CLINICAL TRIAL: NCT06648642
Title: An Open-label Clinical Trial of IR-TMS for AUD and Development of a Neurobiological Biomarker for Craving and Relapse Validated Using a Direct Biochemical Biomarker (Phosphatidylethanol) of Alcohol Use
Brief Title: Image-guided, Robot Navigated Transcranial Magnetic Stimulation (IR-TMS) for Alcohol Use Disorder (AUD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Wellcome Leap Inc. (Industry)
Responsible Party: Principal Investigator, Brett Ginsburg, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000467
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder
Keywords: Transcranial magnetic stimulation; TMS; Phosphatidylethanol
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: A 3-arm open label, adaptive randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Left dorsolateral prefrontal cortex (L-DLPFC) IR-TMS (Active Comparator): Stimulation will be delivered to the L-DLPFC at a depth corrected intensity of 80-95 V/m, using a theta burst stimulation protocol which delivers 1,800 pulses/session. Sessions will be compressed and delivered up to 4 times per day, over the course of 2 weeks.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Dorsomedial prefrontal cortex (DMPFC) IR-TMS (Active Comparator): Stimulation will be delivered to either the DMPFC at a depth corrected intensity of 80-95 V/m, using a theta burst stimulation protocol which delivers 1,800 pulses/session. Sessions will be compressed and delivered up to 4 times per day, over the course of 2 weeks.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Orbitofrontal cortex (OFC) IR-TMS (Active Comparator): Stimulation will be delivered to either the OFC at a depth corrected intensity of 80-95 V/m, using a theta burst stimulation protocol which delivers 1,800 pulses/session. Sessions will be compressed and delivered up to 4 times per day, over the course of 2 weeks.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — TMS applies a strong (~2 Tesla), rapidly changing electro-magnetic field at the scalp to induce electrical current flow in underlying brain tissues
  Other Names: Image-guided, robot-navigated transcranial magnetic stimulation (IR-TMS)

SUMMARY:
This study is testing a new treatment called IR-TMS (image-guided, robot navigated transcranial magnetic stimulation) to see if it can help people who drink too much alcohol to reduce the amount they drink. Participants will be placed into one of three groups, each receiving a slightly different version of this treatment. The study involves going through a few sessions of IR-TMS, having brain scans (MRI), providing blood and urine samples, and answering questions about their drinking and mental health. These activities are part of the study and aren't usually part of regular treatment for alcohol use.

IR-TMS is different from regular treatments like therapy or medication because it uses magnetic fields to target specific parts of the brain. The goal is to see if this treatment can help reduce the urge to drink. There are other options, like sticking with therapy or medication, which are less intense but have been used for a longer time.

DETAILED DESCRIPTION:
Participants with AUD will undergo accelerated IR-TMS treatments and longitudinal fMRI scanning to determine treatment effects and durability. Participants will be recruited and randomized to 1 of 3 treatment target site regions: 1) Left dorsolateral prefrontal cortex; 2) Dorsomedial prefrontal cortex; or 3) Orbitofrontal Cortex. Each participant's target site region will be determined by personalized fMRI connectivity maps. Participants will receive up to 4 IR-TMS treatments per day for up to 10 days (total = 40 accelerated IR-TMS treatments) in an open-label clinical trial with an adaptive treatment design-if one target site region demonstrates superior treatment responses, the remaining participant sample will undergo IR-TMS treatments on that target site.

ELIGIBILITY:
Inclusion Criteria:

1. Two self-reported heavy drinking episodes (>4 drinks for men, >3 for women) or >13 drinks in the last 14 days (at screening)
2. PEth >20 ng/mL (at baseline)
3. Diagnosis of a current, moderate to severe AUD assessed by the The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) substance use checklist
4. Able to attend all study appointments
5. Fluent in English

Exclusion Criteria:

1. Current diagnosis of a moderate or severe substance use disorder (SUD; other than AUD, cannabis, or nicotine)
2. Inability to provide informed consent
3. Alcohol withdrawal-related seizure or hospitalization in the prior 12 months
4. Currently enrolled in AUD treatment
5. Psychiatrically or medically unsafe to participate due to a documented diagnostic history of bipolar disorder, schizophrenia or schizoaffective disorder
6. Any history or signs of serious medical or neurological illness including seizure disorders
7. History of traumatic brain injury (TBI) with loss of consciousness for 20 minutes or more
8. Liver enzymes that are more than 5x the normal range
9. Females will be excluded if they are pregnant
10. Any history or signs of metal objects in the body deemed unsafe for Magnetic Resonance Imaging (MRI) or that may adversely affect image quality of the brain region (e.g. surgical clips, cardiac pacemakers, metal implants, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Measure of Phosphatidylethanol (PEth) level | Baseline, 1 month and 6 months
  Determine if accelerated IR-TMS significantly changes alcohol consumption (as measured by phosphatidylethanol (PEth)) in participants with AUD.

SECONDARY OUTCOMES:
Brain functional connectivity | Baseline to 6 months
  Unified Structural Equation Modeling (SEM) analyses will be used for image analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Brett C Ginsburg, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Be Well Institute, University of Texas Health Science Center - Department of Psychiatry & Behavioral Sciences, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Final copies of all publications, abstracts, and presentations will be archived in the study's repository and made accessible to all study personnel, including the submitted version and any subsequent revisions.
  Public policy will focus on ensuring that all dissemination of research findings from this study is conducted in an accurate, transparent and ethical manner.
Supporting Information: Study Protocol, SAP
Time Frame: At the time of study completion and publication in a peer review journal